CLINICAL TRIAL: NCT07286487
Title: Effects of Glycyrrhetinic Acid on Human Skin in an Acute Irritant Contact Dermatitis Model
Brief Title: Glycyrrhetinic Acid and Acute Irritant Dermatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2181-198-03-04-25-0072; IP-UNIST-35 (Other Grant/Funding Number: Funded by the European Union - NextGenerationEU)
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Irritant Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Irritant | interventions — Glycyrrhetinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- No Treatment and Intact skin (Other): No topical product will be applied. Intact skin.
  Interventions: Other: No Treatment
- Placebo and Intact skin (Placebo Comparator): Topical placebo formulation identical in appearance and vehicle composition to the active preparation but without glycyrrhetinic acid. Used to control for vehicle effects on skin parameters. Intact skin.
  Interventions: Other: Placebo
- Glycyrrhetinic Acid (lower dose) and Intact skin (Experimental): Topical formulation containing a lower concentration of 18β-glycyrrhetinic acid. Designed to evaluate the dose-dependent effect of the active compound on intact skin parameters. Intact skin.
  Interventions: Other: Lower Dose Glycyrrhetinic Acid
- Glycyrrhetinic Acid (higher dose) and Intact skin (Experimental): Topical formulation containing a higher concentration of 18β-glycyrrhetinic acid. Used to assess whether a higher dose enhances anti-inflammatory and barrier-restoring effects compared with the lower dose and placebo.
  Interventions: Other: Higher Dose Glycyrrhetinic Acid
- No Treatment and Irritation (Other): No topical product will be applied. SLS induced skin irritation.
  Interventions: Procedure: SLS induced irritation; Other: No Treatment
- Placebo and Irritation (Placebo Comparator): Topical placebo formulation identical in appearance and vehicle composition to the active preparation but without glycyrrhetinic acid. Used to control for vehicle effects on skin parameters. SLS induced skin irritation.
  Interventions: Procedure: SLS induced irritation; Other: Placebo
- Glycyrrhetinic Acid (lower dose) and Irritation (Experimental): Topical formulation containing a lower concentration of 18β-glycyrrhetinic acid. Designed to evaluate the dose-dependent effect of the active compound on skin recovery and barrier function after irritation. SLS induced skin irritation.
  Interventions: Procedure: SLS induced irritation; Other: Lower Dose Glycyrrhetinic Acid
- Glycyrrhetinic Acid (higher dose) and Irritation (Experimental): Topical formulation containing a higher concentration of 18β-glycyrrhetinic acid. Used to assess whether a higher dose enhances anti-inflammatory and barrier-restoring effects compared with the lower dose and placebo. SLS induced skin irritation
  Interventions: Procedure: SLS induced irritation; Other: Higher Dose Glycyrrhetinic Acid

INTERVENTIONS:
Procedure: SLS induced irritation — Skin irritation will be induced on 4 defined test sites on one forearm (randomly selected forearm) using 60 uL of 1% w/v sodium lauryl sulfate (SLS) aqueous solution under occlusion for a defined period to create a controlled model of acute irritant dermatitis.
  The contralateral forearm will remain untreated and serve as intact skin for comparison.
  Following the induction phase, all test products (placebo and active formulations) will be applied to both irritated and intact sites according to the treatment allocation.
  Arms: Glycyrrhetinic Acid (higher dose) and Irritation; Glycyrrhetinic Acid (lower dose) and Irritation; No Treatment and Irritation; Placebo and Irritation
Other: No Treatment — Designated test area with no topical application after irritation (on the irritated forearm) and on corresponding intact skin (on the non-irritated forearm). Serves as a baseline reference for spontaneous recovery and physiological skin variability.
  Arms: No Treatment and Intact skin; No Treatment and Irritation
Other: Placebo — Topical formulation identical in composition to the active preparations but without glycyrrhetinic acid.
  Used to evaluate the effect of the formulation vehicle on skin parameters. Applied daily to designated test sites on both irritated and intact forearm areas for the duration of the study.
  Arms: Placebo and Intact skin; Placebo and Irritation
Other: Lower Dose Glycyrrhetinic Acid — Topical formulation containing a lower concentration of 18β-glycyrrhetinic acid.
  Designed to assess the effects of the active compound at a lower dose on skin barrier recovery and skin parameters following SLS-induced irritation.
  Applied daily to designated test sites on both irritated and intact forearm areas for the duration of the study.
  Arms: Glycyrrhetinic Acid (lower dose) and Intact skin; Glycyrrhetinic Acid (lower dose) and Irritation
Other: Higher Dose Glycyrrhetinic Acid — Topical formulation containing a higher concentration of 18β-glycyrrhetinic acid.
  Designed to assess the effects of the active compound at a lower dose on skin barrier recovery and skin parameters following SLS-induced irritation.
  Applied daily to designated test sites on both irritated and intact forearm areas for the duration of the study.
  Arms: Glycyrrhetinic Acid (higher dose) and Intact skin; Glycyrrhetinic Acid (higher dose) and Irritation

SUMMARY:
Irritant dermatitis is one of the most common inflammatory skin disorders, caused by exposure to external substances that induce inflammation and immune activation. Standard management includes avoidance of irritants, restoration of the skin barrier using emollients, and the application of anti-inflammatory drugs such as topical corticosteroids. However, due to the risks associated with long-term corticosteroid use, there is an interest in developing emollient formulations enriched with bioactive compounds possessing anti-inflammatory properties. Among those promising compounds is glycyrrhetinic acid.

18β-Glycyrrhetinic acid, a bioactive component of licorice root extract, exhibits potent anti-inflammatory and antioxidant effects. Topical application has demonstrated beneficial outcomes in conditions such as atopic dermatitis, acne, pruritus, and UVB-induced skin damage. Its proposed mechanisms of action include inhibition of key inflammatory enzymes (COX, 5-LOX, iNOS) and promotion of skin regeneration through stimulation of aquaporin-3 expression and enhancement of epidermal turnover.

Topical application of formulations containing 18β-glycyrrhetinic acid will improve skin parameter disturbances caused by irritation induced with sodium lauryl sulfate.

This study aims to evaluate the effects of 18β-glycyrrhetinic acid on human skin parameters in an acute irritant dermatitis model induced by sodium lauryl sulfate, providing further insight into its potential role as an anti-inflammatory and barrier-restoring agent.

Funding:

Funded by the European Union - NextGenerationEU. Views and opinions expressed are however those of the author(s) only and do not necessarily reflect those of the European Union or the European Commission. Neither the European Union nor the European Commission can be held responsible for them.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants aged 18 years or older, of any sex.
* Intact, healthy skin at the test sites.
* No use of systemic or topical corticosteroids, immunomodulators, or antihistamines within the previous three months.
* No use of topical emollients on the test sites within the previous seven days.

Exclusion Criteria:

* Pregnant women, women suspected of being pregnant, and breastfeeding women.
* Non-compliance with the study protocol.
* Voluntary withdrawal or personal decision not to continue participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Transepidermal water loss | Baseline, Irritation Assessment, 3rd, 6th, 8th and 10th day of the treatment
  Tewameter will be used to assess skin barrier function as a measurement of the water loss (g/m2/h).
Hydration | Baseline, Irritation Assessment, 3rd, 6th, 8th and 10th day of the treatment
  Corneometer will be used to estimate skin dryness. It is a relative measurement and uses arbitrary units (AU).
Erythema | Baseline, Irritation Assessment, 3rd, 6th, 8th and 10th day of the treatment
  Mexameter will be used to assess erythema. It is a relative measurement and uses arbitrary units (AU).
Skin elasticity | Baseline, Irritation Assessment, 3rd, 6th, 8th and 10th day of the treatment
  Cutometer will be used to assess skin elasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scheinman PL, Vocanson M, Thyssen JP, Johansen JD, Nixon RL, Dear K, Botto NC, Morot J, Goldminz AM. Contact dermatitis. Nat Rev Dis Primers. 2021 May 27;7(1):38. doi: 10.1038/s41572-021-00271-4. PMID 34045488
- [Background] Johansen JD, Bonefeld CM, Schwensen JFB, Thyssen JP, Uter W. Novel insights into contact dermatitis. J Allergy Clin Immunol. 2022 Apr;149(4):1162-1171. doi: 10.1016/j.jaci.2022.02.002. Epub 2022 Feb 18. PMID 35183605
- [Background] Kang SY, Um JY, Chung BY, Lee SY, Park JS, Kim JC, Park CW, Kim HO. Moisturizer in Patients with Inflammatory Skin Diseases. Medicina (Kaunas). 2022 Jul 1;58(7):888. doi: 10.3390/medicina58070888. PMID 35888607
- [Background] Weisshaar E. Chronic Hand Eczema. Am J Clin Dermatol. 2024 Nov;25(6):909-926. doi: 10.1007/s40257-024-00890-z. Epub 2024 Sep 19. PMID 39300011
- [Background] Kowalska A, Kalinowska-Lis U. 18beta-Glycyrrhetinic acid: its core biological properties and dermatological applications. Int J Cosmet Sci. 2019 Aug;41(4):325-331. doi: 10.1111/ics.12548. Epub 2019 Jun 28. PMID 31166601